CLINICAL TRIAL: NCT05056792
Title: Effects of Plyometric Training vs. Isometric Strengthening of Quadriceps on Strength, Sprint Test, and Single-Leg Triple Hop Test in Soccer Players
Brief Title: Efficacy of Plyometric Training Isometric Strength Training on Quadriceps Strength and Functional Performance.
Acronym: Isometric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Majmaah University (Other)
Responsible Party: Principal Investigator, Shahnaz Hasan, PhD, Associate Professor, Majmaah University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DSR Majmaah University
Record Dates: First submitted 2021-09-14; First posted 2021-09-27 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2021-09

CONDITIONS: Football Players
Keywords: Strength Resisted sprint training; Plyometric training; Function performance; Resisted sprint training
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider
Masking Description: Randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants in this group will receive isometric strength training. (Experimental): Isometric strength training of the quadriceps femoris muscle for 8 weeks.
  Interventions: Other: Isometric strength training for 8 week; Other: Conventional training
- Participants in this group will receive plyometric training. (Sham Comparator): Participants in this group will receive plyometric training for 8 weeks.
  Interventions: Other: Isometric strength training for 8 week; Other: Conventional training

INTERVENTIONS:
Other: Isometric strength training for 8 week — Plyometric training for 8 week
  Other Names: plyometric training training
Other: Conventional training — Conventional training for 8 week

SUMMARY:
This study aims to investigate the influence of an eight-week plyometric and quadriceps strength training program on muscular strength, sprint, and functional performance in collegiate football players.

DETAILED DESCRIPTION:
Sixty collegiate football players aged 18-25 years were recruited, at the university campus. All of them were randomly divided into two experimental and control groups that participated in training for six weeks on alternate days (i.e., three sessions per week), and one control group (n=30) did not train. The control group was instructed to maintain regular activities and avoid any strenuous physical activity during the study.

Under the Declaration of Helsinki, participants were informed about the study's possible risks and benefits, and all participants signed informed consent before participation in the study. The ethical sub-committee of the College of applied medical science, Majmaah, Saudi Arabia approved this study (Ethics Number: MUREC-Jan. 25/COM-2021 / 19-5).

ELIGIBILITY:
Inclusion Criteria:

• Young players aged between 18 and 25 years required frequent sprinting

Exclusion Criteria:

* Current injury to the lower limb.
* Surgery affecting lower limb function.
* Any cardio-respiratory diseases.
* Impairments of the spine or lower extremities.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2021-01-30 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-28 (Actual)

PRIMARY OUTCOMES:
Maximal Voluntary Isometric Contraction Strength (STN) | After 8 weeks of intervention
  Pretest and post intervention strength measure.
Sprint Test (ST) | After 8 weeks of intervention
  Pretest and post intervention sprint measure.
Single-Leg Triple Hop Test (SLTH) | After 8 weeks of intervention
  Pretest and post intervention single-leg triple hop measure.

CONTACTS AND LOCATIONS:
Overall Officials: Shahnaz Hasan, PhD, Principal Investigator — Majmaah University
Locations (1):
- Physiotherapy and Rehabilitation center, Al Majma'ah, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Data has been kept secure with the principal investigator Dr. Shahnaz Hasan due to confidentiality issues.